CLINICAL TRIAL: NCT06954818
Title: A Randomized, Observer-blind, Placebo-controlled, Adaptive Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of SYS6017(a Zoster mRNA Vaccine) in Healthy Participants Aged 40 Years or More
Brief Title: Safety and Immunogenicity of SYS6017 in Healthy Participants Aged 40 Years or More
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SYS6017-001
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Intervention Model Description: The participants are to be randomly assigned to the investigational vaccine or the placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Investigational vaccine of Dosage A (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Investigational vaccine of Dosage B (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Investigational vaccine of Dosage C (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Investigational vaccine of Dosage D (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Investigational vaccine of Dosage E (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: A zoster mRNA vaccine SYS6017 — SYS6017 is an investigational lipid nanoparticle (LNP)-coated mRNA vaccine encoding the glycoprotein E (gE) of VZV, and indicated for active immunization for the prevention of zoster caused by the reactivation of latent VZV.
  Arms: Investigational vaccine of Dosage A; Investigational vaccine of Dosage B; Investigational vaccine of Dosage C; Investigational vaccine of Dosage D; Investigational vaccine of Dosage E
Other: Placebo — saline solution
  Arms: Placebo

SUMMARY:
Herpes zoster is caused by the reactivation of latent varicella-zoster virus (VZV) which stays in latency after its primary infection. Immunosenescence contributes significantly to elevating morbidity associated with aging. Vaccination plays a key role in reducing the disease burden of zoster and the associated complications. This randomized, observer-blind, placebo-controlled, adaptive phase 1 trial aims to evaluate the safety and immunogenicity of an investigational zoster mRNA vaccine in healthy participants aged 40 years or more.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy participants aged 40 years or more;
* 2. Be able to understand the study procedures and comply with the requirements of the protocol for the scheduled visits, voluntarily consent to participate in the study and sign the informed consent form (ICF);
* 3. Being in good health at the discretion of investigators based on medical history inquiry, physical examination, laboratory test and electrocardiograph examination;
* 4. For female participants of childbearing potential: no sexual activity or used effective contraceptive methods within one menstrual cycle before enrollment; no pregnancy plans and agree to used effective contraceptive methods with 8 months after enrollment.

Exclusion Criteria:

* 1. History of zoster;
* 2. History of vaccination with varicella vaccine or zoster vaccine (including investigational vaccine);
* 3. Axillary temperature ≥ 37.1℃ on the day of enrollment or within 24 h before enrollment;
* 4. Have abnormal test or examination result that is of Grade 1 (inclusive) or more in accordance with the Guidelines for Adverse Event Grading Standards for Clinical Trials of Preventive Vaccines (2019) issued by China National Medical Products Administration or other applicable adverse event grading standards referred in the protocol;
* 5. History of allergy to any component of the investigational vaccine, or history of severe allergic reaction (including but not limited to anaphylaxis, allergic laryngeal edema, Henoch-Schonlein purpura, thrombocytopenia purpura or Arthus reaction) to vaccines or medicines;
* 6. History of myocarditis, pericarditis, or idiopathic cardiomyopathy, or any condition that would increase the risk of myocarditis or pericarditis;
* 7. History of demyelinating diseases, including but not limited to Guillain-Barré syndrome, multiple sclerosis, ophthalmoneuromyelitis, acute disseminated encephalomyelitis, etc.
* 8. Current epilepsy or convulsion, severe neurological or psychiatric disorders;
* 9. Have contraindications to intramuscular injection, e.g., diagnosed thrombocytopenia, any coagulation disorders, or current treatment with anticoagulants, etc;
* 10. Active malignant tumor, malignant tumor without adequate treatment, malignant tumor with a potential risk of recurrence during the study;
* 11. Active, unstable, severe or uncontrolled cardiovascular and cerebrovascular diseases, thrombotic diseases, blood and lymphatic system diseases, liver and kidney diseases, respiratory diseases, metabolic diseases, musculoskeletal diseases, autoimmune diseases, etc;
* 12. Have diagnosed immunocompromise or immunosuppression, congenital or functional asplenia, or splenectomy;
* 13. Have received immunosuppressants, immunostimulants, or other immunomodulatory medicines (e.g., corticosteroids, ≥ 20 mg/d prednisone or equivalent) for a long time (defined as 14 days or more), within 6 months before enrollment, or planning to receive the aforementioned medicines during the study; inhaled and topical steroids are allowed;
* 14. Have received whole blood, plasma, serum, immunoglobulins, or monoclonal antibodies within 3 months before enrollment, or planning to receive these products during the study;
* 15. Blood donation or blood loss ≥ 450 mL within 1 month before enrollment, or planning to donate blood during the study;
* 16. Have received any other vaccine within 30 days before enrollment, or planning to receive any other vaccine within 30 days after the last dose;
* 17. Currently participating in or planning to participate in other clinical trials during the study;
* 18. For female participant of childbearing potential: having positive urine pregnancy test, being in pregnancy or lactation before enrollment;
* 19. Unable to comply with the study procedures or adhere to the study requirements, or there are other conditions that make the participation in this study inappropriate, as determined by the investigators.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
solicited adverse events | within 14 days post each vaccination
unsolicited adverse events | within 30 days post each vaccination

SECONDARY OUTCOMES:
serious adverse events | from the first vaccination through 12 months post the second vaccination
adverse events of special interest | from the first vaccination through 12 months post the second vaccination
pregnancy events | from the first vaccination through 12 months post the second vaccination
anti-gE antibody geometric mean concentration, geometric mean fold increase and seroconversion rate. | before the second vaccination, 14 and 30 days post the second vaccination
anti-VZV antibody geometric mean titer, geometric mean fold increase and seroconversion rate. | before the second vaccination, 14 and 30 days post the second vaccination